CLINICAL TRIAL: NCT06416280
Title: Inter-observer Reliability of the Assessment of the Risk of Developing a Venous Thromboembolic Event, the TRiP(Cast) Score, in Patients With Trauma to a Lower Limb Requiring Immobilisation
Brief Title: Inter-observer Reliability of the TRiP(Cast) Score in Patients With Trauma to a Lower Limb Requiring Immobilisation
Acronym: CCASTING
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 24_0131
Record Dates: First submitted 2024-05-06; First posted 2024-05-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism; Thromboprophylaxis; Lower Limb Trauma; Immobilisation Syndrome
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of the TRiP(cast) score — In patients presenting to the emergency department with trauma to a lower limb, the TRiP(cast) score is assessed in accordance with the recommendations. If the patient does not object. The attending physician will then be asked to fill in his implicit assessment of the risk of venous thromboembolism on a paper CRF and then to complete his assessment of the TRiP(cast) score. He will then be free to decide whether or not to anticoagulate the patient.
  At the same time, a doctor not involved in the patient's care will assess the TRiP(cast) score and record it on a paper CRF. The second doctor's assessment will be independent and will have no impact on the patient's management.
  The CRFs will then be analysed and stored. Data will be anonymised during data collection and each patient will be assigned an anonymity number.

SUMMARY:
The aim of the study isto evaluate the inter-observer reliability of the assessment of venous thromboembolic risk using the TRiP(cast) score in patients presenting with trauma to a lower limb requiring immobilisation, and of the clinicians' assessment using the physician's implicit probability (gestalt) compared with the use of the TRiP(cast) score.

DETAILED DESCRIPTION:
Trauma to the lower limbs requiring orthopedic immobilisation (plaster cast or splint) is a frequent reason for seeking emergency care. Because of the venous stasis caused by immobilisation, hypercoagulability and vascular lesions induced by the trauma, these patients are at risk of developing a venous thromboembolic event (VTE). This risk is estimated at around 2% (95% CI 1.3 to 2.7). To reduce the risk of thrombosis, preventive anticoagulants, mainly low molecular weight heparins (LMWH) and fondaparinux, have been shown to be beneficial. However, not all patients have the same thromboembolic risk factors. A targeted strategy should therefore be used to avoid prescribing treatment to low-risk patients and to prescribe it to the sub-group of patients at high risk. The TRiP(cast) score has been developed and validated for this purpose.

In the CASTING study (randomised stepped-wedge trial), patients not receiving thromboprophylaxis on the basis of a TRiP(cast) score <7 had a 3-month rate of symptomatic thromboembolic events of 0.70% (95% CI: 0.21-1.17). Use of the TRiP(cast) score reduced the rate of anticoagulation prescriptions by 26% (24.5% versus 50.4%) without increasing the rate of thromboembolic events at 3 months. Since this study, French recommendations concerning the prescription of anticoagulation treatments have been updated.

Since this study, French recommendations concerning the prescription of preventive anticoagulant treatment have been updated by the SFMU (French Society of Emergency Medicine) and the SFMV (French Society of Vascular Medicine). They were presented in June 2023 and are now applied in all emergency facilities. During the review for the publication of the CASTING study, it was discussed whether it would be useful to evaluate the reliability of this score.

However, the reliability of the measurement and the reproducibility of the score have never been assessed. Given the importance of assessing the risk of venous thromboembolism in patients with lower-limb trauma when deciding whether or not to prescribe thromboprophylaxis, this assessment is essential.

Although this score appears to be objective, there are still items where interpretation may be different. For example, the type of immobilisation cannot be transposed perfectly to all existing immobilisation methods. This study will also be carried out in other European countries. The types of immobilisation vary considerably from one country to another, and the interpretation of certain items could be different. The interpretation of patient characteristics may also vary.

Furthermore, this score has never been compared with the clinician's implicit "gestalt" probability, which is used to define patients at risk of venous thromboembolic events.

It is a real challenge when implementing scores to assess their added value compared with clinical intuition. The use of scores has an initial educational objective, but it is important to know whether clinical intuition would be sufficient to assess this venous thromboembolic risk.

The aim of the study is to evaluate the inter-observer reliability of the assessment of venous thromboembolic risk using the TRiP(cast) score in patients presenting with trauma to a lower limb requiring immobilisation, and of the clinicians' assessment using the physician's implicit probability (gestalt) compared with the use of the TRiP(cast) score.

ELIGIBILITY:
Inclusion Criteria:

* Consultation in one of the emergency departments participating in the study,
* Isolated trauma to a lower limb,
* Rigid immobilisation (plaster or resin) or semi-rigid immobilisation for an expected duration of at least 7 days,
* Patient over 18 years of age,
* Patient affiliated to or benefiting from a social security scheme,
* Patients who have signed a prior informed consent form

Exclusion Criteria:

* Patient taking anticoagulant treatment at the time of the trauma,
* Trauma requiring hospitalisation for more than 48 hours,
* Pregnant, breast-feeding or parturient patients,
* Patient deprived of liberty by judicial or administrative decision,
* Patient under compulsory psychiatric care,
* Patient under legal protection,
* Patients unable to give their free and informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Emergency department patients
Sampling Method: Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary aim is to assess the inter-observer reliability of venous thromboembolic risk assessment using the TRiP(cast) score in patients with lower limb trauma requiring immobilisation. | Day 0
  Outcome measure : The rate of agreement or "concordance" will be estimated by the Kappa coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Delphine DOUILLET, Principal Investigator — University Hospital, Angers
Locations (1):
- DOUILLET Delphine, Angers, France

IPD SHARING:
Plan to Share IPD: No